CLINICAL TRIAL: NCT01836718
Title: An Assessment of Intrahepatic HCV RNA Levels at the Time of Liver Transplantation in Patients With HCV Receiving Antiviral Therapy While on the Liver Transplant Waiting List Compared to Those Not Currently Receiving Therapy
Brief Title: Assessment of Intrahepatic Hepatitis C Virus (HCV) RNA Levels at the Time of Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Schiano, Thomas D., MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: MISP-50064; 13-00099 (Other: Mount Sinai PPHS)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Hepatitis C Virus; Liver Transplantation
Keywords: Hepatitis C Virus; Liver Transplantation; Antiviral Therapy; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, liver explant tissue and hilar lymph nodes will be obtained for testing. With subject consent, any unused specimens will be retained indefinitely for use in future research either related or unrelated to this study, which may include genetic testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HCV RNA (-) on anti-viral therapy: Patients undergoing liver transplantation who are documented HCV viral load undetectable while on antiviral therapy
- HCV RNA (+) on anti-viral therapy: Patients undergoing liver transplantation who are receiving anti-viral therapy and who have a documented detectable HCV viral load
- HCV RNA (+) not on anti-viral therapy: Patients undergoing liver transplantation who are not currently receiving anti-viral therapy and are documented viral load positive will be included and serve as a comparison group

SUMMARY:
The purpose of this study is to measure intrahepatic HCV RNA levels at the time of liver transplantation in patients receiving antiviral therapy while on the liver transplant waiting list. This will eventually be correlated with the degree of hepatic fibrosis present within different geographic sites in the cirrhotic liver. Tissue samples will be obtained from the patient's liver explant as well as hilar lymph nodes. Upon the removal of the cirrhotic liver at the time of transplantation, the explant will be biopsied multiple times in different segments of the liver and preserved for viral detection studies as well as analysis of the degree of fibrosis. Peripheral blood mononuclear cells (PBMCs) will be obtained for viral detection at the time of transplantation. Serum HCV RNA levels will also be obtained at 1 month, 3 months and 6 months post liver transplantation.

Study Hypotheses:

* Virological relapse or non-response is higher is patients with cirrhosis due to failure of antiviral medication to concentrate adequately in a fibrotic liver having an altered sinusoidal micro-architecture
* HCV may persist in different geographic regions of the fibrotic liver in part predicated on blood supply to that area and this may have an effect on overall virological response. These differences in viral persistence and detection may exist in different lobes of the liver or even within a few centimeters within the same portion of the liver parenchyma.
* PBMC and hilar lymph nodes may be extrahepatic reservoirs of HCV viral persistence in patients receiving antiviral therapy and may account for virological relapse post-therapy
* There may be varying degrees of fibrosis within the same cirrhotic liver which may impact on hepatic synthetic function and antiviral response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-80 with chronic HCV on the liver transplant waiting list may be eligible for participation
* The following subjects will be enrolled:

  * Patients undergoing liver transplantation who are documented HCV viral load undetectable while on antiviral therapy
  * Patients receiving anti-viral therapy and who have a detectable HCV viral load
  * Patients not currently receiving antiviral therapy and are HCV PCR (+) will be included and serve as a comparison group

Exclusion Criteria:

* Patients who are co-infected with HIV and/or HBV will not be included

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Hepatitis C on the Mount Sinai Recanati/Miller Transplantation Institute's Liver Transplant Waiting list may be eligible for participation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
HCV RNA PCR levels | Time of Transplantation
  The primary objective is to detect and quantitate HCV RNA PCR levels in different anatomic regions of the liver at the time of liver transplantation to ascertain whether there is similar geographic presence and/or clearance of HCV during antiviral therapy

SECONDARY OUTCOMES:
HCV persistence | Time of Transplantation
  To ascertain whether HCV persistence within the liver is predictive of virological relapse post liver transplantation.
Hepatic Fibrosis | Time of Transplantation
  To assess the degree of hepatic fibrosis at the site of intrahepatic HCV viral detection in order to ascertain whether HCV viral detection correlates with the degree of fibrosis. This study will also examine whether there can be different degrees of hepatic fibrosis in different geographic portions of the same liver and whether there would be a correlation with the patients' natural MELD score, degree of hepatic synthetic function and ultimate virological response to antiviral therapy.
Extrahepatic reservoirs | Time of Transplantation
  To examine whether hilar lymph nodes and PBMC are extrahepatic reservoirs of HCV in patients receiving antiviral therapy and then to correlate this with intrahepatic detection of HCV and overall virological response.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Schiano, MD, Principal Investigator — Mount Sinai School of Medicine Recanati/Miller Transplantation Institute
Locations (1):
- Mount Sinai School of Medicine Recanati/Miller Transplantation Institute, New York, New York, United States